CLINICAL TRIAL: NCT03116451
Title: Nurses' Foot Health and Work Well-being - Development and Testing of an Electronic Foot Health Program
Brief Title: Nurses' Foot Health and Work Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Finnish Work Environment Fund (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Minna Stolt, Principal Investigator, University of Turku
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116464
Record Dates: First submitted 2017-04-05; First posted 2017-04-17 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Foot; Nurses
Keywords: foot health; nurses; work well-being

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot Health Promoting Program (Experimental): The experimental group will receive an electronic intervention (Foot Health Promotion Program, FHPP) for 8 weeks consisting of foot self-care guidance (skin and nail self-care), foot exercises, foot stretching and professional footwear guidance. Each topic includes lectures (delivered via Adobe Presenter) and self-directed learning where participant will go through a list of links to websites and watch videos about foot self-care. In addition, the learning will be evaluated using four individual tasks related to foot self-care.
  Interventions: Behavioral: Foot Health Promoting Program
- Comparison group (No Intervention): The comparison group will not receive any instructions or guidance for foot self-care but participant in the comparison group will complete the same measurement points than experimental group. After the study, the comparison group will also receive the same intervention than experimental group (if effective).

INTERVENTIONS:
Behavioral: Foot Health Promoting Program — An electronic intervention for 8 weeks consisting of foot self-care guidance targeted to nurses.
  Other Names: FHPP
  Arms: Foot Health Promoting Program

SUMMARY:
This study supports and promotes work well-being of nursing personnel from the perspective of foot health in health care organizations. Half of the participants will receive an electronic foot health education program to improve their foot self-care knowledge, while the other will receive anything. The outcomes of this project include recommendations and tested educational program to occupational health care for improving foot health of nurses.

DETAILED DESCRIPTION:
An electronic Foot Health Promoting Program (FHPP) will be tested with nurses using quasi-experimental study design.

The participants will be assigned to experimental (N=130) and comparison (N=130) groups. The experimental group will receive an electronic intervention (Foot Health Promotion Program) for 8 weeks consisting of foot self-care guidance (skin and nail self-care), foot exercises, foot stretching and professional footwear guidance. Detailed components of the intervention will be produced on the bases of survey (part 1) results. The intervention (Figure 3) will be electronic via internet (Moodle platform) where a material package of foot health care will be delivered. Each participant will receive a user account to platform. The platform is divided into four main themes all related to foot health. Each theme consists of two topics of foot health. Each topic includes lectures (delivered via Adobe Presenter) and self-directed learning where participant will go through a list of links to websites (will be evaluated with certain criteria beforehand) and watch videos about foot self-care. In addition, the learning will be evaluated using four individual tasks related to foot self-care. By responding to task a participant will receive an example of the correct answer and using that he/she can evaluate own response and learn by that. Participants' use of different links (quantity) and their paths in the intervention platform will be calculated and analysed. The participants will be tested before the intervention (baseline) and one month (follow-up 1) and four (follow-up 2) months after the intervention. The primary outcome is foot health knowledge and secondary outcomes are foot health, musculoskeletal problems, work ability, health-related quality of life and work satisfaction. Hypothesis is: Increasing nurses' knowledge about foot health will improve their foot health and work ability. Ultimate goal is to develop tools for the occupational health care and improve the attention paid to feet as part of the work ability among nurses.

ELIGIBILITY:
Inclusion Criteria:

* nurses (registered nurses, licensed practical nurses, public health nurses) working in the operating theatre

Exclusion Criteria:

* other health care professionals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Foot self-care knowledge at 4 and 12 weeks | baseline, 4 weeks, 12 weeks
  Measured with Foot Self-Care Knowledge Questionnaire including 11 questions using a "true," "false," or "don't know" response options.

SECONDARY OUTCOMES:
Change from Baseline Foot health at 4 and 12 weeks | baseline, 4 weeks, 12 weeks
  Self-reported foot health questionnaire (SFHQ) will be modified for this study. It will measure self-reported foot health consisting of five subscales: skin, nails, foot structure, foot pain and professional footwear.
Change from Baseline Musculoskeletal Disorders at 4 and 12 weeks | baseline, 4 weeks, 12 weeks
  Nordic Questionnaire measures musculoskeletal disorders in neck, shoulders, upper back, elbows, low back, wrists/hands, hips/thighs, knees and ankles/feet.
Change from Baseline Foot health Status at 4 and 12 weeks | baseline, 4 weeks, 12 weeks
  Foot Health Status Questionnaire measures foot health related to quality of life. There are 4 subscales: foot pain (4 questions), foot function (4 questions), footwear (3 questions), and general foot health (2 questions).
Change from Baseline Work Ability Score at 4 and 12 weeks | baseline, 4 weeks, 12 weeks
  Work Ability Score, assesses workers self-assessed work ability (one item with 0-10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Minna Stolt, PhD, Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stolt M, Katajisto J, Peltonen J, Suhonen R, Leino-Kilpi H. Development and testing of a new electronic foot health promotion programme on nurses' foot self-care. BMC Nurs. 2020 Apr 19;19:29. doi: 10.1186/s12912-020-00423-z. eCollection 2020. PMID 32327936